CLINICAL TRIAL: NCT00868894
Title: A Randomized, Double-masked, Placebo- and Active-controlled, Multi-Center, Dose Escalation Trial of DE-104 Ophthalmic Solution in Japanese and Non-Japanese Subjects With Primary Open-angle Glaucoma or Ocular Hypertension
Brief Title: Safety and Efficacy Study of DE-104 Ophthalmic Solution to Treat Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27-003
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: DE-104 medium concentration
- 2 (Experimental)
  Interventions: Drug: DE-104 high concentration
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo
- 4 (Active Comparator)
  Interventions: Drug: 0.005% latanoprost

INTERVENTIONS:
Drug: DE-104 medium concentration — Topical ocular application
  Arms: 1
Drug: DE-104 high concentration — Topical ocular application
  Arms: 2
Drug: Placebo — Topical ocular application
  Arms: 3
Drug: 0.005% latanoprost — Topical ocular application
  Arms: 4

SUMMARY:
To investigate safety, efficacy, and the dose-response relationship of DE-104 in lowering intraocular pressure in Japanese and Non-Japanese subjects with primary open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Provided signed, written informed consent.
* 18 years of age and older.
* Diagnosed with primary open-angle glaucoma or ocular hypertension.
* If a subject is a female of childbearing potential she must utilize reliable contraceptive throughout the study, and must have a negative urine pregnancy test prior to enrollment into this study.

Exclusion Criteria:

* Females who are pregnant, nursing or planning a pregnancy, or females of childbearing potential who are not using a reliable method of contraception.
* Presence of any abnormality or significant illness that could be expected to interfere with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-03; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To compare the safety and efficacy of two concentrations of DE-104 ophthalmic solution with placebo and 0.005% latanoprost in Japanese and Non-Japanese subjects with primary open-angle glaucoma or ocular hypertension. | 15 days

SECONDARY OUTCOMES:
To investigate the dose-response relationship of DE-104 in lowering intraocular pressure in Japanese and Non-Japanese subjects with primary open-angle glaucoma or ocular hypertension. | 15 days

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Artesia, California
  - Pasadena, California
  - San Francisco, California
  - Honolulu, Hawaii
  - Kailua, Hawaii
  - New York, New York